CLINICAL TRIAL: NCT00631631
Title: Liposomal Muramyl Tripeptide Phosphatidyl Ethanolamine (L-MTP-PE) for High-risk Osteosarcoma
Brief Title: Mifamurtide (L-MTP-PE) for High-Risk Osteosarcoma
Status: Completed | Type: Observational
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MTP-OS-403
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Osteosarcoma
Keywords: Drug Therapy
MeSH Terms: conditions — Osteosarcoma | interventions — mifamurtide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mifamurtide (L-MTP-PE): Mifamurtide (L-MTP-PE), intravenous, at a dose of 2 mg/m^2 twice weekly (at least 3 days apart) for 12 weeks, and then weekly for an additional 24 weeks, for a total of 48 doses in 36 weeks.
  Interventions: Drug: Mifamurtide (L-MTP-PE)

INTERVENTIONS:
Drug: Mifamurtide (L-MTP-PE) — Solution for intravenous infusion
  Other Names: Liposomal Muramyl Tripeptide Phosphatidyl Ethanolamine

SUMMARY:
The purpose of this study was to collect information regarding the safety and tolerability of mifamurtide (liposomal muramyl tripeptide phosphatidyl ethanolamine; L-MTP-PE).

DETAILED DESCRIPTION:
The drug being tested in this study is called mifamurtide (L-MTP-PE; liposomal muramyl tripeptide phosphatidyl ethanolamine). Mifamurtide is being used to treat people with osteosarcoma, a form of cancer.

This was a patient-access study that looked at adverse events, disease progression, and overall survival in study participants.

The study enrolled 205 patients, of whom 204 were treated with mifamurtide intravenously at a dose of 2 mg/m2 twice weekly (at least 3 days apart) for 12 weeks, and then weekly for an additional 24 weeks, for a total of 48 doses in 36 weeks (following surgery for primary or metastatic disease).

This study was conducted in the United States. Participants could receive treatment for up to 9 months. This study was previously mis-categorized as an interventional study.

ELIGIBILITY:
Inclusion Criteria:

1. Had signed informed consent/assent. Voluntary participation in the pharmacokinetic portion of the compassionate access protocol was included in the informed consent but not required for compassionate use participation.
2. Had diagnosis of high grade osteosarcoma with relapsed or recurrent disease, locally or metastatic, with disease not completely resectable or who were unable to complete recommended chemotherapy due to toxicity: relapse, recurrence local or metastatic; unable to have standard surgical resection; abbreviated chemotherapy regimen secondary to toxicity (e.g. hypophosphatemia from ifosfamide, cardiotoxicity from doxorubicin, renal dysfunction from methotrexate, ifosfamide, or cisplatin.)
3. Aged 2 ≤ 50 years.
4. Had adequate hematopoietic function as demonstrated by: 1) Absolute Neutrophil Count (ANC) > 750/microL; Hemoglobin (Hb) > 8 g/dL; Platelets > 30,000/microL.
5. Had adequate hepatic function as documented by 1) ALT < 2.5 x upper limit of normal (ULN) for age; 2) total bilirubin ≤ 1.5 x ULN for age.
6. Had adequate renal function as demonstrated by: 1) Creatinine clearance or radioisotope glomerular filtration rate > 70 mL/min/1.73 m^2; OR, 2) Serum creatinine ≤ 2x ULN for age.
7. Had absence of concurrent active acute infection (i.e., afebrile).
8. In females of child bearing potential (not menopausal for 12 months or no previous surgical sterilization), had a negative pregnancy test. All sexually active participants used an effective means of contraception. Such means included oral contraceptives, Lupron Depot, DepoProvera, and condom with diaphragm and spermicidal jelly.
9. Performance status: Lansky 50-100% (≤ 16 years of age); OR, Eastern Cooperative Oncology Group (ECOG) 0-2 or Karnofsky 50-100% (>16 years of age).

Exclusion Criteria:

1. Had chronic use of corticosteroids or other immunosuppressive agents.
2. Was pregnant or breast-feeding.

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Had diagnosis of high grade osteosarcoma with relapsed or recurrent disease, locally or metastatic, with disease not completely resectable or who were unable to complete recommended chemotherapy due to toxicity: relapse, recurrence local or metastatic; unable to have standard surgical resection; abbreviated chemotherapy regimen secondary to toxicity.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2008-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 12 months or disease progression, whichever occurs first

SECONDARY OUTCOMES:
Serum concentration-time profiles of free and total mifamurtide in 15-20 patients | Just before the start of the first infusion of mifamurtide and at 0.5, 1, 2, 4, 6 and, 24 hours following the start of the first infusion and just prior to the 2nd dose of mifamurtide
Overall survival | From date of enrollment to date of death
Progression-free survival | From date of enrollment to date of first documented disease progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Peter M. Anderson, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - U.T.M.D. Anderson Cancer Center, Houston, Texas